CLINICAL TRIAL: NCT01816334
Title: Safety and Efficacy of Nonsteroidal Antiinflammatory Drug and Glucocorticoids in Acute Sciatica
Brief Title: Safety and Efficacy of Nonsteroidal Antiinflammatory (NSAI)Drug and Glucocorticoids in Acute Sciatica
Acronym: TéAGS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1201
Record Dates: First submitted 2013-03-14; First posted 2013-03-22 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Sciatica
Keywords: sciatica; Anti-Inflammatory Agents, Non-Steroidal; Glucocorticoids
MeSH Terms: conditions — Sciatica | interventions — Methylprednisolone; Ketoprofen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- methylprednisolone (Active Comparator): administration of 60 mg of methylprednisolone at 8:00 am and 100 ml of 0.9 % sodium chloride (placebo) at 6:00 pm
  Interventions: Drug: methylprednisolone; Drug: Sodium Chloride
- Ketoprofen (Active Comparator): administration of 100 mg of ketoprofen at 8:00 am and at 6:00 pm
  Interventions: Drug: Ketoprofen
- sodium chloride (Placebo Comparator): administration of 100 ml of 0.9% sodium chloride (placebo) at 8:00 am and at 6:00 pm
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: methylprednisolone
  Arms: methylprednisolone
Drug: Ketoprofen
  Arms: Ketoprofen
Drug: Sodium Chloride
  Arms: methylprednisolone; sodium chloride

SUMMARY:
The purpose of this study is to determine whether anti-inflammatory drugs or glucocorticoids are effective in the treatment of acute sciatica

ELIGIBILITY:
Inclusion Criteria:

* sciatica <8 weeks resistant to all treatments in ambulatory
* Acute low back pain> 48 hours;
* Non-deficit patients;
* Initial VAS> 40/100;
* Consent of patient
* Conflict disco-radicular concordance with the clinical computed tomography scan or magnetic resonance imaging.
* No of contraindications to methylprednisolone, ketoprofen;
* No registration to another protocol;

Exclusion Criteria:

* Pregnant, parturient, lactating mother;
* Diabetic patient;
* Patient with syndrome from narrowing of the lumbar vertebral canal
* Patient with a history of lumbar surgery <1 year;
* Patient with a Cauda equina syndrome or major motor disability;
* Crural neuralgia
* Patient with a deficit;
* Suspicion of sciatica secondary, ie not conflict-related disco-root: infectious neuritis, fracture on spinal bone tumor ...

associated treatment or pathology contra-indicating administration methylprednisolone, ketoprofen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mean visual analogue scale (VAS) for leg pain (radicular pain) in 3 groups | From day 0 to day 5
  VAS is measured in millimiters (0 to 100). This pain score is recommended in rheumatologic units in France.

SECONDARY OUTCOMES:
Mean visual analogue scale (VAS) for back pain in 3 groups | From day 0 to day 5
  VAS is measured in millimeters (0 to 100).
Assess drug compliance | From day 0 to day 5
  Drug compliance is estimated based on the proportion of the treatment actually administered.
The effect of treatment on the EIFEL Questionnaire | At baseline, 1 and 3 months after intervention
  The EIFEL questionnaire is the translation of the Roland Morris Disability Questionnaire (RMDQ) and has been validated in acute low back pain.
Improvement in Lasegue's sign compared to baseline | At baseline, Day 1,2,3,4 and 5 of study period
  Lasegue's sign is the lumbar pain experienced by the patient on passive movement of the legs during flexion of hip joint i.e. passive straight leg raising. It is assessed as either 'Positive' or 'Negative' sign.
Assess Schober's test | From Day 0 to Day 5
  Schober's test is a test used in rheumatology to measure the ability of patient to flex their lower back
Analgesic consumption | At baseline, day 0, 1, 2, 3, 4 and day 5, 1 and 3 months
  Analgesic consumption between active treatment group and placebo group was registered and differences between groups were calculated and presented as percentual differences.
Surgery or lumbar epidural injection | At 1 and 3 months after intervention
  Number of patient having surgery and/or lumbar epidural injection during study period
Clinical tolerance: adverse events and/or high blood pressure | at baseline, day 1, 2 3, 4 and 5
  Number of adverse events and/or high blood pressure between intervention group.
Biological tolerance | at baseline, day 3 and 5
  measures of leukocytes, erythrocytes, hemoglobin, platelets, serum sodium, potassium, glucose, plasma creatinine between intervention group
Glycemic levels | at baseline, day 1 to 5
  monitoring of glycemic status is measured for each day of treatment
Number of days of hospitalisation sick leave, number of days lost to illness | At baseline, 1 and 3 months
  To assess the cost of sciatica for society

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Hôpital Sud, Échirolles
  - CH d'Uriage, Uriage-les-Bains

REFERENCES:
- [Background] Roncoroni C, Baillet A, Durand M, Gaudin P, Juvin R. Efficacy and tolerance of systemic steroids in sciatica: a systematic review and meta-analysis. Rheumatology (Oxford). 2011 Sep;50(9):1603-11. doi: 10.1093/rheumatology/ker151. Epub 2011 Apr 27. PMID 21525139
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Medications for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):505-14. doi: 10.7326/0003-4819-147-7-200710020-00008. PMID 17909211
- [Background] Vroomen PC, de Krom MC, Slofstra PD, Knottnerus JA. Conservative treatment of sciatica: a systematic review. J Spinal Disord. 2000 Dec;13(6):463-9. doi: 10.1097/00002517-200012000-00001. PMID 11132976
- [Background] Koes BW, Scholten RJ, Mens JM, Bouter LM. Efficacy of non-steroidal anti-inflammatory drugs for low back pain: a systematic review of randomised clinical trials. Ann Rheum Dis. 1997 Apr;56(4):214-23. doi: 10.1136/ard.56.4.214. PMID 9165992
- [Background] Luijsterburg PA, Verhagen AP, Ostelo RW, van Os TA, Peul WC, Koes BW. Effectiveness of conservative treatments for the lumbosacral radicular syndrome: a systematic review. Eur Spine J. 2007 Jul;16(7):881-99. doi: 10.1007/s00586-007-0367-1. Epub 2007 Apr 6. PMID 17415595